CLINICAL TRIAL: NCT02867306
Title: A Phase 1 Open-label, Single-sequence, Drug Interaction Study to Evaluate the Pharmacokinetics of ASP1707 and Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Pharmacokinetics of ASP1707 and Methotrexate in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1707-CL-3002; 2016-001192-76 (EudraCT Number)
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: methotrexate (MTX); Pharmacokinetics; ASP1707; Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — opigolix; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP1707 and methotrexate (MTX) (Experimental): On day 1 patients will receive prescribed dose of MTX. On Days 3 through 8, patients will receive ASP1707 (twice daily). On Day 9, patients will receive a single dose in the morning. A single dose of MTX will be coadministered on Day 8.
  Interventions: Drug: ASP1707; Drug: methotrexate (MTX)

INTERVENTIONS:
Drug: ASP1707 — Oral
Drug: methotrexate (MTX) — Oral

SUMMARY:
The primary purpose of the study is to evaluate the effect of ASP1707 twice daily on the pharmacokinetics of once weekly oral methotrexate (MTX).

This study will also evaluate the effect of MTX on multiple-dose pharmacokinetics of ASP1707, as well as safety and tolerability of coadministration of ASP1707 and MTX in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Patients will check into the clinic on Day -1 and remain in the clinic until all exit procedures have been performed on the morning of Day 10.

ELIGIBILITY:
Inclusion Criteria:

* Female patient must either:

  * Be of nonchildbearing potential: postmenopausal (defined as at least 2 years after last regular menstrual cycle) prior to screening and follicle-stimulating hormone (FSH) ≥ 30 IU/mL, or
  * documented surgically sterile
* Or, if of childbearing potential,

  * Agree not to try to become pregnant during the study and for 28 days or 5 half-lives, whichever is longer, after the final study drug administration;
  * and have a negative urine pregnancy test at screening;
  * and, if heterosexually active, agree to consistently use 2 forms of highly effective birth control (at least one of which must be a barrier method) starting at screening and throughout the study period and for 28 days or 5 half-lives, whichever is longer, after the final study drug administration.
* Male patient and his female spouse/partner who is of childbearing potential must be using highly effective forms of contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continue throughout the study period and for 60 days after the final study drug administration.
* Female patient must agree not to breastfeed starting at screening and throughout the study period, and for 28 days or 5 half-lives, whichever is longer, after the final study drug administration.
* Female patient must not donate ova starting at screening and throughout the study period, and for 28 days or 5 half-lives, whichever is longer, after the final study drug administration.
* Male patient must not donate sperm starting at screening and throughout the study period, and for 60 days after the final study drug administration.
* Patient agrees not to participate in another interventional study while on treatment.
* Patient has a body mass index (BMI) of ≤ 35 kg/m2, inclusive, and must weigh at least 50 kg at screening.
* Patient must have a clinical diagnosis of RA according to the 2010 criteria of the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) at least 6 months prior to screening.
* Patient meets the ACR 1991 revised criteria for RA Global Functional Status I or II.
* Patient must be on concomitant MTX at a stable 10 to 25 mg/week dose for ≥ 28 days prior to day 1 and throughout the study.
* Patient on other medications (excluding MTX) for the treatment or RA at the time of screening must be able to discontinue these medications 28 days or 5 half-lives (whichever is longer) before first study drug dose:

  o Hydroxychloroquine, cyclosporine, leflunomide and sulfasalazine
* Patient use of nonsteroidal anti-inflammatory drugs (NSAIDs), COX-2 inhibitors, folic acid, low dose opioids, hormone replacement therapy (HRT), corticosteroids (prednisone equivalent of ≤ 5 mg/day) for treatment of RA may be allowed in the study. These medications must be stable for ≥ 28 days prior to screening and patients should remain on their regimen throughout the study. Occasional acetaminophen use (less than 2 g/day) may be allowed.
* Patient use of conventional and biologic disease-modifying antirheumatic drugs (DMARDs) used to treat RA may be allowed in this study. These medications must be stable for 4 weeks prior to the study and remain stable during the study. Prior approval for its use must be obtained from the sponsor.

Exclusion Criteria:

* Patient has a previous history of clinically significant systemic disease which might confound the results of the study or pose an additional risk in administering study drug(s) to the patient. This may include, but not be limited to, a history of drug or food allergies, uncompensated heart failure, uncontrolled diabetes mellitus, severe hepatic failure, severe pulmonary disease, or history of mental disease.
* Patient has a history of any malignancy in the past 5 years, except for adequately-treated nonmelanoma skin cancer and adequately-treated-in-situ cervical cancer.
* Patient has a positive serology test for hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) 1+2 antibodies.
* Patient received any breast cancer resistance protein (BCRP) transporter inhibitors or substrates, with the exception of MTX, within 28 days or 5 half-lives, whichever is longer, prior to day 1.
* Patient with liver enzyme test abnormalities, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin > 2 times the upper limit of normal (ULN).
* Patient has a recent history (within the last 6 months) of drug or alcohol abuse (as defined by the Investigator) or a positive urine screen for alcohol or drugs of abuse/illegal drugs at screening or check-in.
* Patient has participated in a previous clinical study with treatment with ASP1707.
* Patient has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to day 1.
* Patient has had any significant blood loss, donated 1 unit (450 mL) of blood, or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day 1.
* Patient is an employee of the Astellas group or vendors involved with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of methotrexate (MTX) in plasma: AUCinf | Up to Day 8
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf)
Pharmacokinetics of methotrexate (MTX) in plasma: Cmax | Up to Day 8
  Maximum concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics of methotrexate (MTX) in plasma: AUClast | Up to Day 8
  Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast)
Pharmacokinetics of methotrexate (MTX) in plasma: tmax | Up to Day 8
  Time after dosing when Cmax occurs (tmax)
Pharmacokinetics of methotrexate (MTX) in plasma: t 1/2 | Up to Day 8
  Apparent terminal elimination half-life (t 1/2)
Pharmacokinetics of methotrexate (MTX) in plasma: CL/F | Up to Day 8
  Apparent total systemic clearance after single or multiple extra-vascular dosing (CL/F)
Pharmacokinetics of methotrexate (MTX) in plasma: Vz/F | Up to Day 8
  Apparent volume of distribution during the terminal elimination phase (Vz/F)
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in plasma: AUClast | Up to Day 8
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in plasma: tmax | Up to Day 8
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in plasma: t 1/2 | Up to Day 8
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in plasma: MPR | Up to Day 8
  Metabolite to parent ratio of AUC using AUC(corr) for the metabolite (corrected by molecular weight ratio of parent to metabolite) (MPR)
Pharmacokinetics of methotrexate (MTX) in urine: Aelast | Up to Day 8
  Cumulative amount of analyte excreted into the urine up to the collection time of the last measurable concentration (Aelast)
Pharmacokinetics of methotrexate (MTX) in urine: Aelast% | Up to Day 8
  Percent of drug dose excreted into urine, feces or bile (Aelast) from time of dosing up to the collection time of the last measurable concentration (Aelast%)
Pharmacokinetics of methotrexate (MTX) in urine: CLR | Up to Day 8
  Renal clearance (CLR)
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in urine: Aelast | Up to Day 8
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in urine: Aelast% | Up to Day 8
Pharmacokinetics of 7-hydroxymethotrexate (7-OH-MTX) in urine: CLR | Up to Day 8
Pharmacokinetics of ASP1707 in plasma: AUCtau | Up to Day 8
  Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau)
Pharmacokinetics of ASP1707 in plasma: Cmax | Up to Day 8
Pharmacokinetics of ASP1707 in plasma: tmax | Up to Day 8
Pharmacokinetics of ASP1707 in plasma: CL/F | Up to Day 8
Pharmacokinetics of ASP1707 in plasma: Ctrough | Up to Day 9
  Concentration immediately prior to dosing at multiple dosing (Ctrough)
Pharmacokinetics of ASP1707 in plasma: MPR | Up to Day 8
Pharmacokinetics of AS1948006 in plasma: AUCtau | Up to Day 8
Pharmacokinetics of AS1948006 in plasma: Cmax | Up to Day 8
Pharmacokinetics of AS1948006 in plasma: tmax | Up to Day 8
Pharmacokinetics of AS1948006 in plasma: Ctrough | Up to Day 8
Pharmacokinetics of AS1948006 in plasma: MPR | Up to Day 8
Safety as assessed by Adverse Events (AEs) | Up to Day 13
Safety assessed by Laboratory Test: hematology | Up to Day 13
Safety assessed by Laboratory Test: biochemistry | Up to Day 13
Safety assessed by Laboratory Test: serology | Up to Day 13
Safety assessed by Laboratory Test: urinalysis | Up to Day 13
Safety assessed by 12- lead electrocardiogram (ECG) | Up to Day 10
  All ECGs should be recorded using the clinic's calibrated equipment. This overall conclusion will be recorded as normal, abnormal not clinically significant, or abnormal clinically significant.
Number of participants with Physical Examination abnormalities and/or adverse events | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc. (APGD)
Locations (1):
- Site MD37301, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=299